CLINICAL TRIAL: NCT05868681
Title: Evaluation of Proprioception in Patients Treated With Surgical External Ankle Ligament Recontruction for Traumatic Ankle Instability
Acronym: ANKLE-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0012824
Record Dates: First submitted 2018-04-12; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2020-04

CONDITIONS: Ankle Sprains; Instability, Joint
Keywords: Ankle instability; Stabilometry
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Proprioceptive training, which will be carried out 1 session lasting one hour twice per week for 5 weeks using Delos instrument with Riva method
  Interventions: Device: Delos instrument (computerized balance board)
- Control group (No Intervention): Normal physiotherapy performed according to standard protocols.

INTERVENTIONS:
Device: Delos instrument (computerized balance board) — Proprioceptive training using Delos instrument (computerized balance board).
  Static and dynamic evaluation through Delos with the Riva method; Physiatric visit; Clinical scores (AOFAs); Functional scores (SPPB); SF12 satisfaction.
  Arms: Study group

SUMMARY:
The objective of the study is to evaluate post-operatively the postural control through the Delos system with the Riva method of patients already treated surgically of external capsulo-ligament reconstruction due to ankle instability.

DETAILED DESCRIPTION:
The patients will then be divided into two control groups: one group will undergo reconditioning through the Delos system and one group will undergo standard rehabilitation treatment.

Primary outcome: improvement of joint stability and postoperative proprioception after reconditioning with the Delos system.

Secondary outcomes: improvement of performance indicators and reduction of disability and satisfaction and assessment of long-term ankle stability after reconditioning with Delos system.

ELIGIBILITY:
Inclusion Criteria:

* patients already undergoing surgery and with at least 4 months of follow-up;
* patients of both sexes aged between 18-40 years;
* patients who have given their informed written consent to participate in the study;
* patients who have given the willingness to reach the Hospital to carry out the checks.

Exclusion Criteria:

* patients with BMI> 30 kg / m2;
* patients with rheumatoid arthritis;
* patients with chronic inflammatory joint diseases;
* patients with pre-existing deambulation kinematics abnormalities (amputations, neuro- muscular diseases, polio, hip dysplasias);
* patients with Severe arthrosis of the ankle (Kellgren-Lawrence> 3);
* patients with Severe knee arthritis (Kellgren-Lawrence> 3);
* patients with severe postural instability;
* patients with cognitive impairments;
* patients with concomitant neurological diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Static and Dynamic Stability Index | 5 weeks from the start of rehabilitation treatment
  Evaluation of proprioception and mechanical stability of the post-operative ankle undergoing to reconditioning with a Delos device through Static and Dynamic Stability Index.

SECONDARY OUTCOMES:
Personal perception of the patient | 5 weeks from the start of rehabilitation treatment
  Subjective perception of the patient evaluated by administering clinical questionnaires (AOFAS ankle hindfoot)
Clinical test | 5 weeks from the start of rehabilitation treatment
  Stability of the ankle operated evaluated by clinical test

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopedic Institute (IOR), Bologna, Italy

IPD SHARING:
Plan to Share IPD: No